CLINICAL TRIAL: NCT06690255
Title: Trial of an Online Spanish Pivotal Response Treatment Training in Autism Spectrum Disorder (PRT-OS)
Brief Title: Trial of an Online Spanish Pivotal Response Treatment Training in Autism Spectrum Disorder
Acronym: PRT-OS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of California, Santa Barbara (Other)
Responsible Party: Principal Investigator, Grace Gengoux, Clinical Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-77671
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spanish PRT Online (Experimental): Participating parents will receive access to a 12-week online course designed to teach Pivotal Response Treatment (PRT) strategies in Spanish. The course includes 10 instructional lessons and check-ins with a researcher via secure videoconference.
  Interventions: Behavioral: Pivotal Response Treatment

INTERVENTIONS:
Behavioral: Pivotal Response Treatment — PRT will target functional communication abilities

SUMMARY:
The goal of this clinical trial is to understand if an online course in Spanish can help Spanish-speaking parents use Pivotal Response Treatment (PRT) to support language and social skills in young children with Autism Spectrum Disorder (ASD). This study aims to reach families who may have trouble accessing autism services due to language, location, or cost barriers. The main questions it hopes to answer are:

* Can Spanish-speaking parents learn to effectively use PRT techniques to support their child's communication?
* Does this training improve children's language and social interactions?

Researchers will evaluate the effectiveness of the online course for parents who participate in regular virtual check-ins and submit videos showing their practice with PRT.

Participants in the study will:

* Complete online lessons over 12 weeks that teach PRT methods, specifically designed for Spanish-speaking parents
* Meet with a research team member every few weeks by phone or video to ask questions and receive feedback
* Provide video recordings of interactions with their child to track progress
* Complete brief surveys about their experience and child's communication abilities

By focusing on Spanish-speaking families, this study aims to increase access to effective autism support and reduce gaps in care. Researchers hope the findings will help develop better resources for families facing similar barriers and improve language and social outcomes for children with autism.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 to 5 years, 11 months at the time of consent
* Diagnosis of Autism Spectrum Disorder (ASD), confirmed through medical records and/or parent questionnaire
* Significant language delay, indicated by scores 2 standard deviations (SD) below the average for ages 2 and 3, or 3 SD below the average for ages 4 and 5 on the Vineland-3 Communication subscale or Expressive V-scale
* A Spanish-speaking parent or primary caregiver available to consistently participate in study activities and implement PRT in Spanish
* Stable on any psychotropic medications or biomedical interventions for at least 1 month before baseline, with no anticipated changes during the study
* Consistent treatment or intervention services (such as ABA, Floortime, or speech therapy) and stable school placement for at least 1 month before baseline, with no expected changes
* Limited to no more than 60 minutes of one-on-one speech therapy per week

Exclusion Criteria:

* Primary language of the child or parent is not Spanish
* Either the child or parent has a severe psychiatric disorder or an unstable medical condition
* Prior exposure to or adequate trial of Pivotal Response Treatment, resulting in the parent achieving fidelity in PRT implementation at baseline
* The child is currently receiving more than 15 hours of one-on-one Applied Behavior Analysis (ABA) therapy per week

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-12-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in Parent Fidelity of PRT Implementation from Baseline to Week 12 | Baseline, Week 12
  Based on behavioral coding of parent-child interaction videos in the home

SECONDARY OUTCOMES:
Change in Child Frequency of Functional Utterances from Baseline to Week 12 | Baseline, Week 12
  Based on behavioral coding of parent-child interaction videos in the home and parent report measures
Change in Child Frequency of Functional Utterances from Baseline to Week 12 | Baseline, Week 12
  Based on parent-report on the MacArthur-Bates Communicative Development Inventories
Change in Child Socialization and Communication from Baseline to Week 12 | Baseline, Week 12
  Based on clinician-rated Clinical Global Impressions Scale (CGI)
Change in Child Socialization and Communication from Baseline to Week 12 | Baseline, Week 12
  Based on parent-rated Vineland Adaptive Behavior Scale, Third Edition (VABS-3)

IPD SHARING:
Plan to Share IPD: No